CLINICAL TRIAL: NCT03170076
Title: Pattern of Skin Manifestations in Chronic Hepatitis c Virus Patients Before and After Direct Acting Anti Viral Drugs: Prospective Controlled Clinical Trial
Brief Title: Pattern of Skin Manifestations in Chronic Hepatitis c Virus Patients Before and After Direct Acting Anti Viral Drugs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hagar Maher, Dermatologic resident, Assiut University
Other Study IDs: skin manifestations in HCV
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Hepatitis C, Chronic
Keywords: skin manifestations - hepatitis c virus
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* Hepatitis C is an infectious disease caused by the hepatitis C virus (HCV) that primarily affects the liver. It is one of the main causes of chronic liver diseases worldwide .
* According to World Health Organization (WHO), 2011 , Egypt has particularly high rates of Hepatitis C (22%).
* Hepatitis C virus (HCV) is known to induce both hepatic and extra-hepatic manifestations. About 17% of HCV patients present with at least one skin manifestation, which can be directly or indirectly induced by chronic HCV infection .

DETAILED DESCRIPTION:
* Skin diseases which are certainly related with chronic HCV infection are mixed cryoglobulinemia, lichen planus , porphyria cutanea tarda, Chronic pruritus and necrolytic acral erythema; conditions that may share a possible association with HCV infection .
* while several immune-mediated inflammatory skin conditions, such as psoriasis, chronic urticaria and vitiligo, have been only rarely reported in the setting of chronic HCV infection .
* Peginterferon based regimen with or without ribavirin were the mainstay of HCV treatment with a cure rate of about 50%, Although these regimens were lengthy, complex, had significant side-effects and high failure rates .
* They also had higher rate of exacerbated dermatologic conditions such as discoid lupus, psoriasis and Lichen planus .
* Recently, Newer all-oral anti viral drugs regimens began to be approved for use in 2014. These regimens, involve one pill daily for 12 weeks, they have achieved sustained virologic response of over 90% and have more tolerable side effect profiles.
* Recently, The European Association for Study of Liver (EASL) 2015, American Association for the Study of Liver Diseases (AASLD) and Infectious Diseases Society of America (IDSA) have now recommended that all chronically infected HCV patient should be offered treatment with new oral antiviral drugs .

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HCV infection eligible for treatment with new (DAADs) and having:

   A- Normal Complete Blood Count ( hemoglobin not less than 10 gm/dl ). B- Mild to moderate impairment of Liver function test and kidney function test.

   C- Positive polymerase chain reaction for HCV virus. D- Controlled Blood sugar .
2. Patients > 18 years

Exclusion Criteria:

1. Patients on treatment for skin disease.
2. Pregnancy and lactation.
3. Patients <18 years.
4. Patients not eligible for oral anti hepatitis C drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patient are from assiut city
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
local skin examination | three months
  examination of skin manifestations in patients with hepatitis c under treatment with direct acting anti viral drugs

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel P, Malik K, Krishnamurthy K. Cutaneous Adverse Events in Chronic Hepatitis C Patients Treated With New Direct-Acting Antivirals: A Systematic Review and Meta-Analysis. J Cutan Med Surg. 2016 Jan;20(1):58-66. doi: 10.1177/1203475415595775. Epub 2015 Jul 10. PMID 26162860
- [Background] Berk DR, Mallory SB, Keeffe EB, Ahmed A. Dermatologic disorders associated with chronic hepatitis C: effect of interferon therapy. Clin Gastroenterol Hepatol. 2007 Feb;5(2):142-51. doi: 10.1016/j.cgh.2006.06.010. Epub 2006 Aug 17. PMID 16919505
- [Background] Strader DB, Wright T, Thomas DL, Seeff LB; American Association for the Study of Liver Diseases. Diagnosis, management, and treatment of hepatitis C. Hepatology. 2004 Apr;39(4):1147-71. doi: 10.1002/hep.20119. No abstract available. PMID 15057920
- [Background] Cacoub P, Bourliere M, Lubbe J, Dupin N, Buggisch P, Dusheiko G, Hezode C, Picard O, Pujol R, Segaert S, Thio B, Roujeau JC. Dermatological side effects of hepatitis C and its treatment: patient management in the era of direct-acting antivirals. J Hepatol. 2012 Feb;56(2):455-63. doi: 10.1016/j.jhep.2011.08.006. Epub 2011 Aug 30. PMID 21884670